CLINICAL TRIAL: NCT06727032
Title: Validation of an AI Software for Detection of Brain Metastases on MRI: AIDED Versus UNAIDED Performance
Brief Title: Automated Detection of Brain Metastases on MRI
Acronym: BrainMets AI
Status: Enrolling by invitation | Type: Observational
Sponsor: Robovision BV (Industry)
Collaborators: Netherlands Cancer Institute - NKI (Unknown)
Responsible Party: Sponsor
Other Study IDs: CI-2024-BrainMetsAI; IRBd20-090 (Other: IRB NKI-AVL)
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Brain Metastasis AI — There will be no intervention

SUMMARY:
This reader study aims at assessing whether the radiologist aided with AI software has at least a non-inferior performance than without AI assistance in detecting brain metastases.

200 retrospective MRI images will be included in the study with 100 positive and 100 negative exams.

Assessment will be completed by 12 readers with varying level of experience. This is a Retrospective Multiple-Reader Multiple-Case (MRMC) randomised study.

ELIGIBILITY:
Inclusion Criteria:

* subjects older than 18 years with a known or possible primary extracranial cancer who undergo MRI for diagnosis, treatment planning or follow-up of brain metastases.

Exclusion Criteria:

* subjects with primary intracranial tumor(s), with more than 10 brain metastases, with meningeal metastases, with radiation necrosis, or post brain surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Brain Metastasis
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Detection accuracy | 3 months
  Demonstrate that the accuracy for detecting brain metastases by radiologists on MRI using the software (AIDED) is at least non-inferior to that of radiologists not using the software (UNAIDED).

SECONDARY OUTCOMES:
Reading time | 3 months
  Demonstrate that the AIDED radiologists reading time for detecting brain metastases is significantly lower than for UNAIDED radiologists.
Inter-reader agreement | 3 months
  Demonstrate that AIDED reading reduces detection variation between observers/readers in brain metastasis detection.

CONTACTS AND LOCATIONS:
Locations (1):
- Netherlands Cancer Institute, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No